CLINICAL TRIAL: NCT01536561
Title: Phase I Study of Radiolabeled Monoclonal Antibody Anti-B1 for the Treatment of B-Cell Lymphomas
Brief Title: Study of Radiolabeled Monoclonal Antibody Anti-B1 for the Treatment of B-Cell Lymphomas and Extended Study to Determine the Safety and Efficacy of Coulter Clone® 131Iodine-B1 Radioimmunotherapy of Advanced Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 104728
Record Dates: First submitted 2012-01-26; First posted 2012-02-22 (Estimated); Results first posted 2012-03-30 (Estimated); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Lymphoma, Non-Hodgkin
Keywords: Tositumomab and/or Iodine I 131 Tositumomab; B-cell non-Hodgkin's lymphoma; Dose-limiting toxicity; Bexxar
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, B-Cell | interventions — tositumomab I-131

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- open-label, dose escalation (Experimental): Each subject will undergo two phases of study. The first phase, termed "tracer Study", involves the injection of low-radioactivity doses (about 5 mCi) of 131-I anti-B1 for the purposes of determining the rate of whole body clearance of radiation so that a whole body radiation can be calculated. The calculated whole-body radiation dose per mCi administered can then be used to determined how many mCi will be required to deliver a specified whole-body radiation dose in the second phase of the study for each patient, termed radio-immunotherapy dose in a tracer-projected whole-body radiation dose will be used for dose escalation with a minimum of three subjects per dose level.
  Interventions: Biological: Radiolabeled Monoclonal Antibody Anti-B1 for the Treatment of B-Cell Lymphomas (Tositumomab and Iodine I 131 Tositumomab)

INTERVENTIONS:
Biological: Radiolabeled Monoclonal Antibody Anti-B1 for the Treatment of B-Cell Lymphomas (Tositumomab and Iodine I 131 Tositumomab) — 131-I anti-B1 is the product of 131-I labeling of the anti-CD20 murine monoclonal antibody and the anti-B1 antibody itself is an intact IgG2a murine monoclonal antibody which has specificity far the CD20 antigen on human B cells. Anti-B1 is a clear, colorless liquid. 131-I labeling of the anti-B1 antibody will be carried out by iodogen technique. Trace labeling of the antibody will involve the labeling of approximately 1 to 3 mg of antibody with 5 mCi of 131-I.

SUMMARY:
Phase I/II, single-center, dose-escalation study of the safety, pharmacokinetics, dosimetry, and efficacy of TST/I-131 TST for the treatment of patients with chemotherapy-refractory or resistant low-grade, intermediate-grade, or high-grade B-cell lymphoma. Subjects received 1 to 3 dosimetric doses followed by a therapeutic dose of TST/I-131 TST. Study BEX104526 was a follow-up study of the long-term safety and efficacy data from the surviving patients who completed at least 2 years of follow-up following administration of TST/I 131 TST on Study BEX104728.

Dosimetric dose: Subjects received 1 to 3 dosimetric doses of TST/I-131 TST, followed by a therapeutic dose of TST/I-131 TST. Subjects received various doses of unlabeled TST (0, 95 or 475 mg) to determine the dose of unlabeled TST that optimized the radiation dose delivered to the tumor by TST/I-131 TST. The unlabeled TST was followed by 5 milliCurie (mCi) of I-131 TST. Serial whole body sodium iodide scintillation probe counts were obtained daily, for at least 5 days, in order to determine the rate of whole body clearance of radioactivity (residence time). The residence time was used to determine the radioactive clearance for the subject and the activity (in mCi) of I-131 required to deliver the desired TBD of radiation during the therapeutic dose. Because 475 mg was determined to be the optimal pre-dose of TST in the first subjects entered, the last 34 subjects received a single dosimetric dose that was preceded by an infusion of 475 mg of TST.

Therapeutic dose: Groups of 3-6 subjects were enrolled at successively higher whole-body radiation dose levels beginning at a total body dose (TBD) of 25 centiGray (cGy). The TBD of each subsequent dose level was escalated by 10 cGy. Subjects who had undergone bone marrow transplantation (BMT) underwent a separate dose escalation (10 cGy TBD increase per dose level) beginning at a TBD level of 65 cGy. The MTD was defined as the highest dose level at which 0/3 or 1/6 subjects experienced dose-limiting toxicity (DLT). DLT was defined as follows:

Any Grade 4 hematologic toxicity (National Cancer Institute [NCI] criteria) lasting greater than 7 days, or Any Grade 3 hematologic toxicity lasting greater than 2 weeks, or Any Grade 3 or 4 nonhematologic toxicity Redosing. Subjects who achieved tumor regression were considered for re-dosing, using the original therapeutic dose of TST/I-131 TST, at the time the tumor was no longer shrinking in an attempt to upgrade their response.

Retreatment. Subjects who achieved partial (PR) or complete response (CR) were considered for retreatment following relapse of their NHL, if progression occurred ≥6 weeks following the therapeutic dose. The original therapeutic dose of TST/I-131 TST was given unless a grade 2 or greater toxicity had been encountered, in which case a reduced dose was administered for the repeat therapeutic dose.

DETAILED DESCRIPTION:
Phase I/II, single-center, dose-escalation study of the safety, pharmacokinetics, dosimetry, and efficacy of TST/I-131 TST for the treatment of patients with chemotherapy-refractory or resistant low-grade, intermediate-grade, or high-grade B-cell lymphoma. Subjects received 1 to 3 dosimetric doses followed by a therapeutic dose of TST/I-131 TST. Study BEX104526 was a follow-up study of the long-term safety and efficacy data from the surviving patients who completed at least 2 years of follow-up following administration of TST/I 131 TST on Study BEX104728.

Dosimetric dose: Subjects received 1 to 3 dosimetric doses of TST/I-131 TST, followed by a therapeutic dose of TST/I-131 TST. Subjects received various doses of unlabeled TST (0, 95 or 475 mg) to determine the dose of unlabeled TST that optimized the radiation dose delivered to the tumor by TST/I-131 TST. The unlabeled TST was followed by 5 milliCurie (mCi) of I-131 TST. Serial whole body sodium iodide scintillation probe counts were obtained daily, for at least 5 days, in order to determine the rate of whole body clearance of radioactivity (residence time). The residence time was used to determine the radioactive clearance for the subject and the activity (in mCi) of I-131 required to deliver the desired TBD of radiation during the therapeutic dose. Because 475 mg was determined to be the optimal pre-dose of TST in the first subjects entered, the last 34 subjects received a single dosimetric dose that was preceded by an infusion of 475 mg of TST.

Therapeutic dose: Groups of 3-6 subjects were enrolled at successively higher whole-body radiation dose levels beginning at a total body dose (TBD) of 25 centiGray (cGy). The TBD of each subsequent dose level was escalated by 10 cGy. Subjects who had undergone bone marrow transplantation (BMT) underwent a separate dose escalation (10 cGy TBD increase per dose level) beginning at a TBD level of 65 cGy. The MTD was defined as the highest dose level at which 0/3 or 1/6 subjects experienced dose-limiting toxicity (DLT).

DLT was defined as follows:

Any Grade 4 hematologic toxicity (National Cancer Institute [NCI] criteria) lasting greater than 7 days, or Any Grade 3 hematologic toxicity lasting greater than 2 weeks, or Any Grade 3 or 4 nonhematologic toxicity Redosing: Subjects who achieved tumor regression were considered for re-dosing, using the original therapeutic dose of TST/I-131 TST, at the time the tumor was no longer shrinking in an attempt to upgrade their response.

Retreatment: Subjects who achieved a partial response (PR) or complete response (CR) were considered for retreatment following relapse of their NHL, if progression occurred ≥6 weeks following the therapeutic dose. The original therapeutic dose of TST/I-131 TST was given unless a grade 2 or greater toxicity had been encountered, in which case a reduced dose was administered for the repeat therapeutic dose.

Subjects who completed at least 2 years of follow-up in BEX104728 were enrolled in LTFU Study BEX104526 for continued radiographic response evaluations and safety evaluations every 6 months for years 3 through 5 post-treatment and annually for years 6 through 10 post-treatment. Subjects in BEX104526 were assessed for survival and disease status, including subsequent therapy for NHL, and for long-term safety, including the development of hypothyroidism, myelodysplastic syndrome (MDS), acute myelogenous leukemia (AML), and any other secondary malignancies. Additionally, subjects were followed for the development of any adverse event(s) (AEs) deemed by the Principal Investigator as being possibly or probably related to a subject's treatment with TST/I-131 TST. Laboratory evaluations, consisting of thyroid stimulating hormone (TSH) level and complete blood cell count with a differential and platelet count, were obtained annually through year 10 post-treatment.

Study assessments included demographic and baseline characteristics; tumor response, duration of response, survival (progression-free survival [PFS] and overall survival [OS]), adverse events (AEs), incidence of human anti-murine antibody (HAMA), incidence of hypothyroidism, and serious (fatal and non-fatal) adverse events (SAEs).

Dosing;"Dosimetric Doses", Intravenous (IV) administration of unlabeled TST (0, 95 or 475 mg) was administered to determine the dose of unlabeled TST that optimized the radiation dose to the tumor. This was followed by 5 mCi of I-131 TST. Serial whole body sodium iodide scintillation probe counts were obtained daily, for at least 5 days, in order to determine the rate of whole body clearance of radioactivity (residence time). The residence time was used to determine the radioactive clearance from the subject and subsequently the activity (in mCi) of Iodine-131 required to deliver the desired TBD of radiation during the therapeutic dose of TST/I-131 TST. Because 475 mg was determined to be the optimal pre-dose of tositumomab in the first subjects entered, the last 34 subjects received a single dosimetric dose that was preceded by an infusion of 475 mg of tositumomab (Source Data: Listing 13).

"Therapeutic Dose", Groups of 3-6 subjects were treated at successively higher therapeutic whole body radiation doses, beginning at a TBD of 25 cGy. The TBD was escalated in 10 cGy increments in subsequent dose level cohorts until the MTD was achieved. A separate determination of MTD was conducted for subjects who had undergone prior BMT. This was initiated at a TBD of 65 cGy TBD and increased in 10 cGy increments until determination of the MTD. The MTD was defined as the dose at which fewer than 1/3 or 2/6 subjects experienced DLT, i.e. any Grade 4 hematologic toxicity (absolute neutrophil count [ANC], platelets, hemoglobin, white blood count [WBC] lasting > 7 days or any Grade 3 hematologic toxicity lasting > 14 days, as defined in Section 4.1.

Re-Dosing; Subjects who achieved tumor regression were considered for re-dosing, using the original therapeutic dose of TST/I-131 TST, at the time the tumor was no longer shrinking in an attempt to upgrade their response. Patients were not redosed sooner than 6 weeks following a therapeutic dose.

Retreatment (≥6 weeks following therapeutic dose); Subjects who achieved a PR or CR were considered for retreatment following relapse of their NHL. The original therapeutic dose of TST/I-131 TST was given unless a Grade 2 or greater toxicity had been encountered, in which case the dose level immediately below the original dose was administered.

ELIGIBILITY:
Inclusion Criteria

* Subjects had histologically-confirmed NHL.
* Subjects with low-, intermediate-, or high-grade histologies, according to the International Working Formulation.
* Subjects had relapsed after or had failed to respond to at least 1 prior chemotherapy regimen.
* Subjects had evidence that their tumor tissue expressed the CD20 antigen.

Exclusion Criteria

* ≥25% bone marrow involvement.
* Absolute granulocyte count ≥1500 cells/mm3 or platelet count ≤100,000 platelets/mm3.
* Creatinine ≥2.0 mg/dL, bilirubin ≥2.0 mg/dL.
* Cytotoxic chemotherapy, radiation therapy, immunosuppressants, or cytokine treatment within 4 weeks of study entry.
* Active infection, collagen vascular disease, vasculitis, glomerulonephritis, New York Heart Association class II or IV heart disease and/or serious illness.
* Prior external beam radiation therapy such that the maximum tolerated dose level for any normal organ would be exceeded by additional irradiation.
* Pregnancy.
* Allergy to iodine or previous sensitization to mouse protein as documented by positive anti-mouse antibody ELISA test.
* Known brain metastases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 1990-04-24 (Actual); Primary Completion 1997-07-02 (Actual); Study Completion 2009-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Kaminski MS, Estes J, Zasadny KR, Francis IR, Ross CW, Tuck M, Regan D, Fisher S, Gutierrez J, Kroll S, Stagg R, Tidmarsh G, Wahl RL. Radioimmunotherapy with iodine (131)I tositumomab for relapsed or refractory B-cell non-Hodgkin lymphoma: updated results and long-term follow-up of the University of Michigan experience. Blood. 2000 Aug 15;96(4):1259-66. PMID 10942366
- See also: Results for study 104728 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/104728?search=study&search_terms=104728#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 104728 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 104728 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 104728 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 104728 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 104728 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 104728 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 104728 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: After an initial treatment (IT), 14 participants (14 of the 59 particpants receiving the IT) who achieved a partial or complete response and subsequently developed progressive disease were retreated (administered at either the initial dose or a reduced dose if a >=Grade toxicity had occurred after the IT) at the time of disease progression.
Pre-assignment Details: Participants received radioimmunotherapy of tositumomab (TST) and Iodine I 131 TST in 2 phases: Phase 1, dosimetric dose; Phase 2, therapeutic dose. After radioimmunotherapy, participants could have entered a 10-year Long-Term Follow-Up study (Study BEX104526; NCT00240591) for continued evaluation.
Groups:
- TST and Iodine I 131 TST: Participants received 1 to 3 dosimetric doses (DD) consisting of 0, 95, or 475 milligrams (mg) of tositumomab (TST) intravenously (IV) followed by 5.0 millicurie (mCi) of Iodine (I 131) TST IV. This was followed by a therapeutic dose (TD) administered 7-14 days after the DD, starting at a total body dose (TBD) of 25 centiGray (cGy) or 65 cGy (only for participants who had undergone bone marrow transplantation) with increments of 10 cGy at each dose level (DL) until the maximum tolerated dose (MTD) was achieved. Participants were re-dosed with a second TD when their tumor stopped regressing (was no longer shrinking). Participants who had completed at least 2 years of follow-up after administration of TST/I 131 TST during the TD phase and had signed the informed consent to participate in the Long-Term Follow-Up (LTFU) study (BEX104526) were followed for up to 10 years. Participants did not receive any study medication during the LTFU study.
Period: Dosimetric and Therapeutic Treatment
Arm/Group | TST and Iodine I 131 TST
Started | 59
Completed | 0
Not Completed | 59
Not completed — Progressive Disease | 40
Not completed — Received Alternate Treatment | 2
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 1
Not completed — Death | 2
Not completed — Enrolled in Study BEX104526 | 13
Period: Long-Term Follow-Up
Arm/Group | TST and Iodine I 131 TST
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | TST and Iodine I 131 TST
Number analyzed (Participants) | 59
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.9 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 37
Race/Ethnicity, Customized [Number; unit: participants]
  White | 54
  Hispanic | 2
  Black | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants (Par.) During Initial Treatment Exposed to the Indicated Dose Levels of the Therapeutic Dose (TD), Re-dose, and Total Dose (TD + Re-dose)
Description: Par. (groups of 3-6) received the TD at a total body dose (TBD) of 25 centiGray (cGy) or 65 cGy (par. who had bone marrow transplantation), increasing by 10 cGy increments at each dose level, until the maximum tolerated dose (MTD) was achieved. The MTD was defined as the highest dose level at which 0/3 or 1/6 par. experienced dose-limiting toxicity (DLT): any Grade 4 hematologic toxicity (National Cancer Institute criteria) lasting >7 days, any Grade 3 hematologic toxicity lasting >2 weeks, or any Grade 3/4 nonhematologic toxicity. Not Applicable (NA) indicates that no par. were re-dosed.
Time Frame: Participants who completed at least 2 years of follow-up in Study BEX104728 were invited to enroll in BEX104526 for long-term follow-up. Participants were evaluated in Study BEX104728 and Study BEX104526 for up to 15.6 years.
Population: Intent-to-Treat (ITT) Exposed Population: all participants who were enrolled into the study and received at least one dose of study drug.
Measure: Number; unit: participants
Groups:
- TST and Iodine I 131 TST: Initial Treatment: Participants received 1 to 3 dosimetric doses (DD) consisting of 0, 95, or 475 milligrams (mg) of tositumomab (TST) intravenously (IV) followed by 5.0 millicurie (mCi) of Iodine (I 131) TST IV. This was followed by a therapeutic dose (TD) administered 7-14 days after the DD, starting at a total body dose (TBD) of 25 centiGray (cGy) or 65 cGy (only for participants who had undergone bone marrow transplantation) with increments of 10 cGy at each dose level (DL) until the maximum tolerated dose (MTD) was achieved. Participants were re-dosed with a second TD when their tumor stopped regressing (was no longer shrinking). Participants who had completed at least 2 years of follow-up after administration of TST/I 131 TST during the TD phase and had signed the informed consent to participate in the Long-Term Follow-Up (LTFU) study (BEX104526) were followed for up to 10 years. Participants did not receive any study medication during the LTFU study.
Arm/Group | TST and Iodine I 131 TST: Initial Treatment
Number analyzed (Participants) | 59
participants
  TD=0cGy+Re-dose=NA; Total=0cGy | 6
  TD=25cGy+Re-dose=NA; Total=25cGy | 1
  TD=25cGy+Re-dose=25cGy; Total=50cGy | 2
  TD=35cGy+Re-dose=NA; Total=35cGy | 4
  TD=45cGy+Re-dose=NA; Total=45cGy | 8
  TD=45cGy+Re-dose=45cGy; Total=90cGy | 1
  TD=55cGy+Re-dose=NA; Total=55cGy | 8
  TD=65cGy+Re-dose=NA; Total=65cGy | 5
  TD=65cGy+Re-dose=65cGy; Total 130cGy | 1
  TD=75cGy+Re-dose=NA; Total=75cGy | 18
  TD=75cGy+Re-dose=65cGy; Total=140cGy | 1
  TD=75cGy+Re-dose=75cGy; Total=150cGy | 1
  TD=85cGy+Re-dose=NA; Total=85cGy | 3

2. Primary Outcome: Number of Participants During Retreatment Exposed to the Indicated Dose Levels of the TD, Re-dose, and Total Dose (TD + Re-dose)
Description: Retreatment was administered to participants either at the initial TD of TST/I 131 TST or at a reduced dose if a >=Grade 2 toxicity had occurred after initial treatment, until the MTD was achieved. The MTD was defined as the highest dose level at which 0/3 or 1/6 participants experienced DLT: any Grade 4 hematologic toxicity (National Cancer Institute criteria) lasting >7 days, any Grade 3 hematologic toxicity lasting >2 weeks, or any Grade 3/4 nonhematologic toxicity. Not Applicable (NA) indicates that no participants were re-dosed.
Time Frame: as for outcome 1
Population: ITT Exposed Population
Measure: Number; unit: participants
Groups:
- TST and Iodine I 131 TST: Retreatment: After the "Initial Treatment" (DD of TST and Iodine I 131 TST, followed by TD), participants who achieved a partial response (PR:>=50% reduction in the sum of the products of the longest perpendicular diameters of all measurable lesions; no new lesions) or complete response (CR: complete resolution of all disease-related radiological abnormalities and the disappearance of all signs and symptoms related to the disease) and subsequently developed progressive disease were retreated at the time of disease progression. Retreatment was administered either at the initial TD of TST/I 131 TST or at a reduced dose if a Grade 2 or greater toxicity had occurred after the "Initial Treatment." Participants who had completed at least 2 years of follow-up after administration of TST/I 131 TST during the TD phase and had signed the informed consent to participate in the LTFU study (BEX104526) were followed for up to 10 years. Participants did not receive any study medication during the LTFU study.
Arm/Group | TST and Iodine I 131 TST: Retreatment
Number analyzed (Participants) | 14
participants
  TD=25cGy+Re-dose=NA; Total=25cGy | 1
  TD=35cGy+Re-dose=NA; Total=35cGy | 1
  TD=38cGy+Re-dose=NA; Total=38cGy | 2
  TD=45cGy+Re-dose=NA; Total=45cGy | 1
  TD=45cGy+Re-dose=45cGy; Total=90cGy | 1
  TD=55cGy+Re-dose=NA; Total=55cGy | 2
  TD=60cGy+Re-dose=NA; Total=60cGy | 1
  TD=65cGy+Re-dose=NA; Total=65cGy | 2
  TD=75cGy+Re-dose=NA; Total=75cGy | 3

3. Primary Outcome: Maximum Tolerated Dose (MTD) of TST/I 131 TST Evaluated in the Study
Description: Participants who had prior bone marrow transplantation (BMT) initiated TD at 65 cGy TBD, whereas those who had no prior BMT initiated TD at 25 cGy TBD. The MTD was defined as the highest dose level at which 0/3 or 1/6 par. experienced DLT: any Grade 4 hematologic toxicity (National Cancer Institute criteria) lasting >7 days, any Grade 3 hematologic toxicity lasting >2 weeks, or any Grade 3/4 nonhematologic toxicity. Not Applicable (NA) indicates that no par. were re-dosed.
Time Frame: as for outcome 1
Population: ITT Exposed Population
Measure: Number; unit: Total body radiation dose in cGy
Arm/Group | TST and Iodine I 131 TST: Initial Treatment
Number analyzed (Participants) | 59
Total body radiation dose in cGy
  Participants who had not undergone BMT | 75
  Participants who had undergone BMT | 45

4. Primary Outcome: Tumor/Organ Dosimetry of TST/I 131 TST for All Predoses (Initial Treatment)
Description: Serial whole body sodium iodide scintillation probe counts were obtained from participants approximately 1 hour after the administration of the dosimetric dose and then daily for at least 5 days. Gamma camera images of participants were used to calculate the amount of radiation that accumulated in the target tumor and normal organs (tumor/organ dosimetry). Spleen volume may vary based on disease status, and volume correction allows for a comparison of spleen dose across participants.
Time Frame: Serial anterior and posterior gamma whole body scans were obtained 1 hour after the administration of the dosimetric dose (on Day 0), and then daily for at least 5 days until Day 7
Population: ITT Exposed Population. Of the 59 participants analyzed, 23 received 2 or 3 dosimetric doses (DD); tumor/organ dosimetry was calculated for all 86 DD. The "n" in the category title reflects the number of DD, which will differ for each target organ depending on whether adequate gamma camera images were available for analysis after each of the 86 DD.
Measure: Mean (Standard Deviation); unit: cGy/75 cGy TBD
Units Other Than Participants: dosimetric doses
Arm/Group | TST and Iodine I 131 TST: Initial Treatment
Number analyzed (Participants) | 59
Number analyzed (dosimetric doses) | 86
cGy/75 cGy TBD
  Spleen (volume-corrected), n=77 | 477.68 (235.95)
  Tumor (average), n=57 | 1074.27 (704.8)
  Kidney (average), n=46 | 607.57 (185.66)
  Liver (average), n=46 | 261.26 (72.03)
  Lungs (average), n=46 | 192.35 (67.53)
  Urine Bladder Wall (average), n=86 | 242.59 (93.24)
  Bone marrow (average), n=38 | 101.25 (16.10)
  Blood (average), n=42 | 368.60 (96.30)
  Testes (average), n=45 | 58.06 (6.14)
  Ovaries (average), n=20 | 71.03 (4.42)

5. Secondary Outcome: Tumor/Organ Dosimetry at the Indicated Predoses of 475 mg, 95 mg, and 0 mg (Initial Treatment)
Description: The effect of unlabeled TST pre-treatment on targeting of radioactive TST was evaluated. Serial whole body sodium iodide scintillation probe counts were obtained from participants approximately 1 hour after the administration of the dosimetric dose (DD) and then daily for at least 5 days. Initially, participants received either two or three DDs, each of which was preceded by a pre-dose of unlabeled tositumomab (0, 95, or 475 mg) to determine the dose of unlabeled tositumomab that optimized the radiation dose to tumor. The tumor radiation absorbed dose was determined using gamma camera images.
Time Frame: as for outcome 4
Population: ITT Exposed Population. Participants who received unlabelled doses of 0 mg, 95 mg, or 475 mg were analyzed. Of the 59 participants analyzed, 23 received 2 or 3 dosimetric doses (DD); tumor/organ dosimetry was calculated for all 86 DD. The "n" in the category title reflects the number of DD, which will differ for each target organ.
Measure: Mean (Standard Deviation); unit: cGy/75 cGy TBD
Units Other Than Participants: dosimetric doses
Arm/Group | TST and Iodine I 131 TST: Initial Treatment
Number analyzed (Participants) | 59
Number analyzed (dosimetric doses) | 86
cGy/75 cGy TBD
  475 mg Predose, Spleen (volume-corrected); n=36 | 411.5 (217.40)
  475 mg Predose, Tumor (average); n=28 | 1023.04 (711.44)
  95 mg Predose, Spleen (volume-corrected); n=21 | 451.77 (238.40)
  95 mg Predose, Tumor (average); n=14 | 1177.3 (650.3)
  0 mg, Spleen (volume-corrected); n=20 | 624 (210.26)
  0 mg, Tumor (average); n=15 | 1073.75 (776.1)

6. Secondary Outcome: Number of Participants (Par.) With the Indicated Response as Assessed by the Investigator
Description: Par. with response include those with Complete Response (CR: complete resolution of all disease-related radiological abnormalities and the disappearance of all signs and symptoms related to the disease), Clinical Complete Response (CCR: complete resolution of all disease-related symptoms; residual foci, thought to be residual scar tissue, are present), or Partial Response (PR: >=50% reduction in the sum of the products of the longest perpendicular diameters of all measurable lesions; no new lesions).
Time Frame: as for outcome 1
Population: ITT Exposed Population. Only those participants evaluable for response were analyzed.
Measure: Number; unit: participants
Groups:
- TST and Iodine I 131 TST: Retreatment: After the "Initial Treatment" (DD of TST and Iodine I 131 TST, followed by TD), participants who achieved a partial response (PR:>=50% reduction in the sum of the products of the longest perpendicular diameters of all measurable lesions; no new lesions) or complete response (CR: complete resolution of all disease-related radiological abnormalities and the disappearance of all signs and symptoms related to the disease) and subsequently developed progressive disease were retreated at the time of disease progression. Retreatment was administered either at the initial TD of TST/I 131 TST or at a reduced dose if a Grade 2 or greater toxicity had occurred after the "Initial Treatment." Participants who had completed at least 2 years of follow-up after administration of TST/I 131 TST during the TD phase and had signed the informed consent to participate in the LTFU study (BEX104526) were followed for up to 10 years. Participants did not receive any study medication during the LTFU stu
Arm/Group | TST and Iodine I 131 TST: Initial Treatment | TST and Iodine I 131 TST: Retreatment
Number analyzed (Participants) | 57 | 14
participants
  CR | 20 | 4
  CCR | 0 | 0
  PR | 22 | 4

7. Secondary Outcome: Number of Participants (Par.) With Confirmed Response as Assessed by the Investigator
Description: Responses had to be confirmed by 2 separate evaluations occurring >=4 weeks apart. Par. with confirmed response include those with Complete Response (CR: complete resolution of all disease-related radiological abnormalities and the disappearance of all signs and symptoms related to the disease), Clinical Complete Response (CCR: complete resolution of all disease-related symptoms; residual foci, thought to be residual scar tissue, are present), or Partial Response (PR: >=50% reduction in the sum of the products of the longest perpendicular diameters of all measurable lesions; no new lesions).
Time Frame: as for outcome 1
Population: ITT Exposed Population. Only those participants evaluable for confirmed response were analyzed.
Measure: Number; unit: participants
Arm/Group | TST and Iodine I 131 TST: Initial Treatment | TST and Iodine I 131 TST: Retreatment
Number analyzed (Participants) | 44 | 9
participants
  Confirmed CR | 20 | 4
  Confirmed CCR | 0 | 0
  Confirmed PR | 9 | 3

8. Secondary Outcome: Duration of Response for All Unconfirmed Responders (CR, CCR, or PR) as Assessed by the Investigator
Description: Duration of response is defined as the time from the first documented response until disease progression.
Time Frame: as for outcome 1
Population: ITT Exposed Population. Only those participants with unconfirmed response (CR, CCR, or PR) and those who experienced progressive disease were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TST and Iodine I 131 TST: Initial Treatment | TST and Iodine I 131 TST: Retreatment
Number analyzed (Participants) | 42 | 8
months | 8.5 [4.1 to 13.0] | 7.7 [4.4 to 96.5]

9. Secondary Outcome: Time to Progression of Disease or Death
Description: Time to progression or progression-free survival is defined as the time from the dosimetric dose to the first documented occurrence of disease progression or death.
Time Frame: as for outcome 1
Population: ITT Exposed Population. Only those participants who experienced progression were evaluated.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TST and Iodine I 131 TST: Initial Treatment | TST and Iodine I 131 TST: Retreatment
Number analyzed (Participants) | 55 | 14
months | 5.7 [3.4 to 8.3] | 4.9 [1.6 to 12.8]

10. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from the treatment start date to the date of death from any cause.
Time Frame: as for outcome 1
Population: ITT Exposed Population. Only those participants who died during the study and during the follow-up period were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TST and Iodine I 131 TST: Initial Treatment | TST and Iodine I 131 TST: Retreatment
Number analyzed (Participants) | 33 | 12
months | 46.4 [30.0 to 92.8] | 45.0 [7.4 to 103.6]

11. Secondary Outcome: Half-life: Initial Half-life (t1/2 Alpha) and Terminal Half-life (t1/2 Beta) of I 131 TST for the Antibody Predose Levels of 0 mg, 95 mg, and 475 mg
Description: t1/2 alpha is the estimated initial or alpha phase half-life in a two-compartmental pharmacokinetic model . t1/2 beta is the estimated terminal or beta phase half-life in a two-compartmental pharmacokinetic model; also denoted as t1/2. Half-life measures how long it takes for the concentration of drug in the blood to decrease by half.
Time Frame: Blood samples were collected at the end of the infusion (Study Day 0) and at 0.5, 1, 2, 4, 12, 24, 36, 48, 72, 96, and 120 hours following the end of the infusion.
Population: ITT Exposed Population. The sample size ("n") in the category titles is the number of infusions (dosing occasions) with parameter results.
Measure: Mean (Standard Deviation); unit: hours (hr)
Units Other Than Participants: infusions
Arm/Group | TST and Iodine I 131 TST: Initial Treatment
Number analyzed (Participants) | 59
Number analyzed (infusions) | 161
hours (hr)
  0 mg, t1/2 alpha, n=24 | 6.2 (5.7)
  95 mg, t1/2 alpha, n=34 | 6.0 (6.5)
  475 mg, t1/2 alpha, n=96 | 6.7 (6.8)
  0 mg, terminal t1/2 beta, n=24 | 63.2 (51.5)
  95 mg, terminal t1/2 beta, n=35 | 72.6 (41.3)
  475 mg, terminal t1/2 beta, n=102 | 84.5 (52.9)

12. Secondary Outcome: Clearance (CL) of I 131 TST for the Indicated Antibody Predose Levels
Description: Clearance is defined as the volume of blood from which drug is removed per unit time and is a measure of the rate at which drug is removed from the body after the dose.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Milliliters per hour (mL/hr)
Units Other Than Participants: infusions
Arm/Group | TST and Iodine I 131 TST: Initial Treatment
Number analyzed (Participants) | 59
Number analyzed (infusions) | 161
Milliliters per hour (mL/hr)
  0 mg, n=24 | 205 (229)
  95 mg, n=35 | 99.4 (78.4)
  475 mg, n=102 | 72.1 (39.0)

13. Secondary Outcome: Area Under the Concentration Time Curve (AUC) of I 131 TST for the Indicated Antibody Predose Levels
Description: Area under the concentration-time curve from the end of the infusion extrapolated to infinite time. AUC measures how much drug is in the system over time after infusion. ID, injected dose.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: %ID * hours per milliliter (%ID.hr/mL)
Units Other Than Participants: infusions
Arm/Group | TST and Iodine I 131 TST: Initial Treatment
Number analyzed (Participants) | 59
Number analyzed (infusions) | 161
%ID * hours per milliliter (%ID.hr/mL)
  0 mg, n=24 | 0.838 (0.453)
  95 mg, n=35 | 1.42 (0.73)
  475 mg, n=102 | 1.68 (0.74)

14. Secondary Outcome: Maximum Blood Concentration (Cmax) of I 131 TST for the Indicated Antibody Predose Levels
Description: Cmax is defined as the maximum observed concentration of the drug in blood.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: % Injected Dose per milliliter (%ID/mL)
Units Other Than Participants: infusions
Arm/Group | TST and Iodine I 131 TST: Initial Treatment
Number analyzed (Participants) | 59
Number analyzed (infusions) | 161
% Injected Dose per milliliter (%ID/mL)
  0 mg, n=24 | 0.0164 (0.0046)
  95 mg, n=35 | 0.0190 (0.0042)
  475 mg, n=102 | 0.0194 (0.0041)

15. Secondary Outcome: Volume of Distribution at Steady State (Vss) of I 131 TST for the Indicated Antibody Predose Levels
Description: Vss is defined as the volume of distribution of the drug at steady state.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: liters
Units Other Than Participants: infusions
Arm/Group | TST and Iodine I 131 TST: Initial Treatment
Number analyzed (Participants) | 59
Number analyzed (infusions) | 161
liters
  0 mg, n=24 | 13.0 (12.3)
  95 mg, n=35 | 7.74 (4.25)
  475 mg, n=102 | 7.08 (2.16)

16. Secondary Outcome: Number of Participants Who Developed Human Anti-mouse Antibodies (HAMA Postivitiy) After Receiving Tositumomab
Description: Tositumomab is a murine (mouse) antibody (immunoglobulin) of the IgG2a subclass. Participants in this study were evaluated to determine whether they developed an immune response to study treatment, as evident by human anti-mouse antibodies (HAMA) after administration of tositumomab and iodine I 131 tositumomab. A positive HAMA value indicates that the participant developed human anti-mouse antibodies above the HAMA assay threshold, and a negative HAMA value indicates either the absence or a below threshold level of human anti-mouse antibodies.
Time Frame: as for outcome 1
Population: ITT Exposed Population. Only those participants evaluable for HAMA were analyzed.
Measure: Number; unit: participants
Arm/Group | TST and Iodine I 131 TST: Initial Treatment | TST and Iodine I 131 TST: Retreatment
Number analyzed (Participants) | 58 | 4
participants
  Positive | 9 | 2
  Negative | 49 | 2

17. Secondary Outcome: Time to HAMA Positivity From the First Dosimetric Dose (Time From Baseline [Dosimetric Dose] to the First Reported Presence of HAMA)
Description: as for outcome 16
Time Frame: as for outcome 1
Population: ITT Exposed Population. Participants who converted to HAMA positivity were analyzed.
Measure: Median (Full Range); unit: days
Arm/Group | TST and Iodine I 131 TST: Initial Treatment | TST and Iodine I 131 TST: Retreatment
Number analyzed (Participants) | 9 | 2
days | 15.0 [12 to 194] | 1271 [19 to 2523]

18. Secondary Outcome: Number of Participants With the Indicated Type of Infection
Description: An infection is the colonization of a host organism by a parasite species. Infecting parasites seek to use the host's resources to reproduce, often resulting in disease. Specimen samples of the body fluid are cultured for testing whether the infectious organism is present and grown in the culture media to assess the growth pattern of the organisms present in the specimen. The culture results could be positive or negative. The positive culture results indicate that the tested participant has the infection under investigation, in which case therapeutic treatment with anti-infective is required.
Time Frame: as for outcome 1
Population: ITT Exposed Population
Measure: Number; unit: participants
Arm/Group | TST and Iodine I 131 TST: Initial Treatment | TST and Iodine I 131 TST: Retreatment
Number analyzed (Participants) | 59 | 14
participants
  Any Infection; n=59, 14 | 24 | 2
  No Infection; n=59, 14 | 35 | 12
  Upper Respiratory Tract Infection; n=24, 2 | 6 | 1
  Urinary Tract Infection; n=24, 2 | 5 | 1
  Nasopharyngitis; n=24, 2 | 2 | 0
  Respiratory Tract Infection; n=24, 2 | 2 | 0
  Sinusitis; n=24, 2 | 2 | 0
  Device Related Infection; n=24, 2 | 1 | 0
  Eye Infection; n=24, 2 | 1 | 0
  Hemophilus Infection; n=24, 2 | 1 | 0
  Herpes Virus Infection; n=24, 2 | 1 | 0
  Herpes Zoster; n=24, 2 | 1 | 0
  Infusion Site Cellulitis; n=24, 2 | 1 | 0
  Pneumonia; n=24, 2 | 1 | 0
  Pneumonia Streptococcal; n=24, 2 | 1 | 0
  Postoperative Wound Infection; n=24, 2 | 1 | 0
  Staphylococcal Sepsis; n=24, 2 | 1 | 0
  Vestibular Neuronitis; n=24, 2 | 1 | 0
  Viral Infection; n=24, 2 | 1 | 0
  Viral Upper Respiratory Tract Infection; n=24, 2 | 1 | 0
  Sepsis; n=24, 2 | 0 | 1

19. Secondary Outcome: Time to Nadir for the Indicated Hematologic Laboratory Parameters
Description: Nadir is defined as the lowest laboratory value recorded following the administration of the study medication.
Time Frame: as for outcome 1
Population: ITT Exposed Population. Only those participants for which nadir could be calculated were analyzed. Some participants did not have post-baseline data available.
Measure: Median (Full Range); unit: days
Arm/Group | TST and Iodine I 131 TST: Initial Treatment | TST and Iodine I 131 TST: Retreatment
Number analyzed (Participants) | 57 | 14
days
  Time to nadir, ANC, n=40, 12 | 44.5 [8 to 97] | 44.5 [28 to 111]
  Time to nadir, hemoglobin, n=57, 14 | 34.0 [2 to 119] | 49.5 [5 to 111]
  Time to nadir, platelets, n=57, 14 | 34.0 [2 to 97] | 41.0 [23 to 104]
  Time to nadir, WBC count, n=57, 14 | 41.0 [2 to 119] | 48.0 [5 to 100]

20. Secondary Outcome: Time to Recovery to Baseline for the Indicated Hematologic Laboratory Parameters
Description: Time to recovery to baseline is the time required for recovery from nadir values to baseline values.
Time Frame: as for outcome 1
Population: as for outcome 19
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | TST and Iodine I 131 TST: Initial Treatment | TST and Iodine I 131 TST: Retreatment
Number analyzed (Participants) | 46 | 4
days
  Time to recovery to baseline, ANC, n=23, 2 | 79.0 [57.0 to 108.0] | 74.0 [44.0 to 74.0]
  Time to recovery to baseline, hemoglobin, n=46, 4 | 42.0 [34.0 to 55.0] | 38.5 [6.0 to NA] — The SAS procedure was not able to calculate the upper limit of the confidence interval.
  Time to recovery to baseline, platelets, n=45, 4 | 57.0 [48.0 to 76.0] | 39.0 [26.0 to 39.0]
  Time to recovery to baseline, WBC count, n=46, 3 | 69.0 [49.0 to 91.0] | 77.0 [56.0 to 77.0]

21. Secondary Outcome: Nadir Values for the Hematologic Parameters ANC, Platelets, and WBC Count
Description: Nadir is defined as the lowest laboratory value recorded following the administration of study medication. ANC is a measure of the number of neutrophil granulocytes present in the blood. Neutrophils are a type of WBC that fights against infection. Platelets and WBCs are types of blood cells.
Time Frame: as for outcome 1
Population: as for outcome 19
Measure: Median (Full Range); unit: 1000 cells/millimeters cubed (mm^3)
Arm/Group | TST and Iodine I 131 TST: Initial Treatment | TST and Iodine I 131 TST: Retreatment
Number analyzed (Participants) | 57 | 14
1000 cells/millimeters cubed (mm^3)
  ANC, n=40, 12 | 1.0 [0 to 5] | 1.3 [0 to 5]
  Platelets, n=57, 14 | 74.0 [2 to 292] | 79.5 [3 to 224]
  WBC count, n=57, 14 | 2.7 [0 to 9] | 3.3 [1 to 6]

22. Secondary Outcome: Nadir Values for Hemoglobin, a Hematologic Parameter
Description: Nadir is defined as the lowest laboratory value recorded following the administration of study medication. Hemoglobin is the iron-containing oxygen-transport metalloprotein in the red blood cells.
Time Frame: as for outcome 1
Population: ITT Exposed Population
Measure: Median (Full Range); unit: G/dL
Arm/Group | TST and Iodine I 131 TST: Initial Treatment | TST and Iodine I 131 TST: Retreatment
Number analyzed (Participants) | 59 | 14
G/dL | 10.9 [6 to 14] | 11.7 [5 to 14]

ADVERSE EVENTS:
Time Frame: Participants who completed at least 2 years of follow-up in Study BEX104728 were invited to enroll in BEX104526 for long-term follow-up. Participants were evaluated in Study BEX104728 and Study BEX104526 for up to 15.6 years.
Arm/Group | TST and Iodine I 131 TST: Initial Treatment | TST and Iodine I 131 TST: Retreatment
Serious Adverse Events (participants affected / at risk) | 17/59 | 7/14
Other Adverse Events (participants affected / at risk) | 55/59 | 12/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TST and Iodine I 131 TST: Initial Treatment (N=59) | TST and Iodine I 131 TST: Retreatment (N=14)
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 5
Acute Myeloid Leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Squamous Cell Carcinoma of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Anal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Carcinoid Tumour Pulmonary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lip and/or Oral Cavity Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Serum Sickness (Immune system disorders) | 2 | 0
Anaphylactic Reaction (Immune system disorders) | 1 | 0
Anaphylactoid Reaction (Immune system disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 3 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 0
Leukopenia (Blood and lymphatic system disorders) | 2 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Hemophilus Infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Pneumonia Streptococcal (Infections and infestations) | 1 | 0
Staphylococcal Sepsis (Infections and infestations) | 1 | 0
Pyrexia (General disorders) | 2 | 0
Fatigue (General disorders) | 1 | 0
Necrotising Panniculitis (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TST and Iodine I 131 TST: Initial Treatment (N=59) | TST and Iodine I 131 TST: Retreatment (N=14)
Pyrexia (General disorders) | 31 | 5
Fatigue (General disorders) | 20 | 3
Chills (General disorders) | 17 | 4
Pain (General disorders) | 2 | 0
Asthenia (General disorders) | 1 | 1
Axillary Pain (General disorders) | 1 | 0
Catheter Site Rash (General disorders) | 1 | 0
Chest Pain (General disorders) | 1 | 0
Ill-Defined Disorder (General disorders) | 1 | 0
Infusion Site Inflammation (General disorders) | 1 | 0
Infusion Site Phlebitis (General disorders) | 1 | 0
Medical Device Complication (General disorders) | 1 | 0
Mucous Membrane Disorder (General disorders) | 1 | 0
Oedema Peripheral (General disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 20 | 7
Vomiting (Gastrointestinal disorders) | 8 | 1
Diarrhea (Gastrointestinal disorders) | 6 | 1
Constipation (Gastrointestinal disorders) | 3 | 0
Gastritis (Gastrointestinal disorders) | 3 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 2 | 1
Abdominal Pain (Gastrointestinal disorders) | 2 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0
Diarrhea Hemorrhagic (Gastrointestinal disorders) | 1 | 0
Fecal Incontinence (Gastrointestinal disorders) | 1 | 0
Paraesthesia Oral (Gastrointestinal disorders) | 1 | 0
White Blood Cells < 2000 cells/cm^3 (Investigations) | 22 | 4
Absolute Neutrophil Count <1000 cells/cm^3 (Investigations) | 21 | 6
Platelets <50000 cells/cm^3 (Investigations) | 18 | 3
Hemoglobin <8.0 g/dL (Investigations) | 11 | 2
Upper Respiratory Tract Infection (Infections and infestations) | 6 | 1
Urinary Tract Infection (Infections and infestations) | 5 | 1
Nasopharyngitis (Infections and infestations) | 2 | 0
Respiratory Tract Infection (Infections and infestations) | 2 | 0
Sinusitis (Infections and infestations) | 2 | 0
Device related infection (Infections and infestations) | 1 | 0
Eye infection (Infections and infestations) | 1 | 0
Herpes Virus Infection (Infections and infestations) | 1 | 0
Herpes Zoster (Infections and infestations) | 1 | 0
Infusion Site Cellulitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Postoperative Wound Infection (Infections and infestations) | 1 | 0
Vestibular Neuronitis (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 1 | 0
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 8 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 1
Erythema (Skin and subcutaneous tissue disorders) | 5 | 0
Rash (Skin and subcutaneous tissue disorders) | 5 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0
Skin Irritation (Skin and subcutaneous tissue disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 2
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 4 | 1
Musculoskeletal Discomfort (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 6 | 3
Dizziness (Nervous system disorders) | 5 | 0
Hypoaesthesia (Nervous system disorders) | 2 | 0
Sciatica (Nervous system disorders) | 1 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal Dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal Ulcer (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 7 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 1 | 0
Diplopia (Eye disorders) | 1 | 0
Eye Irritation (Eye disorders) | 1 | 0
Photophobia (Eye disorders) | 1 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 4 | 1
Oliguria (Renal and urinary disorders) | 1 | 0
Ureteric Obstruction (Renal and urinary disorders) | 1 | 0
Urinary Incontinence (Renal and urinary disorders) | 1 | 0
Urinary Retention (Renal and urinary disorders) | 1 | 1
Bladder Pain (Renal and urinary disorders) | 0 | 1
Flushing (Vascular disorders) | 2 | 0
Hypotension (Vascular disorders) | 2 | 0
Serum Sickness (Immune system disorders) | 2 | 0
Weight Decreased (Investigations) | 2 | 0
Disorientation (Psychiatric disorders) | 1 | 0
Nightmare (Psychiatric disorders) | 1 | 0
Sinus Tachycardia (Cardiac disorders) | 1 | 1
Angina Pectoris (Cardiac disorders) | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Ear Discomfort (Ear and labyrinth disorders) | 0 | 1
Ear Injury (Injury, poisoning and procedural complications) | 0 | 1
Liver Function Test Abnormal (Investigations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.